CLINICAL TRIAL: NCT03306134
Title: The Effect of Beta-blockers in Substance P Levels and the Swallowing Function
Acronym: BETASP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Marta Miarons, Clinical pharmacist, Hospital de Mataró
Other Study IDs: 2017/05
Record Dates: First submitted 2017-09-22; First posted 2017-10-10 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Beta Blockers; Swallowing Disorder; Substance P
MeSH Terms: conditions — Deglutition Disorders | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BETA-BLOCKERS: Patients taking beta-blockers with or without dysphagia
  Interventions: Diagnostic Test: Dysphagia
- NO BETA-BLOCKERS: Patients not taking beta-blockers with or without dysphagia
  Interventions: Diagnostic Test: Dysphagia

INTERVENTIONS:
Diagnostic Test: Dysphagia — An overall assessment is going to be carry out by a multidisciplinary team during the visit.
  Swallowing assessment is going to be performed during the visit. We are going to use: (i) the Eating Assessment Tool (EAT-10), which is a short 10-item, easy to use, self-administered questionnaire [4]. Although the EAT-10 is considered to be predominantly a questionnaire on FHS, some items on HR-QoL are also included. The sum score of this 10-item questionnaire ranges from 0 to 40, and (ii) the Sydney Swallowing Questionnaire (SSQ) to clinically assess the severity of the symptoms of dysphagia, if present.
  All subjects are going to be submitted to the volume-viscosity swallow test (V- VST)
  Other Names: Diagnostic test

SUMMARY:
A non-randomised, prospective study to assess the effects of beta-blockers on substance P levels and the swallowing function. The study is going to be carry out in the Gastrointestinal Physiology Laboratory of the Hospital de Mataró (Spain). All participants will be actively recruited from a Linked hospital and primary care database. We include two groups: the first group (group 1) are participants taking beta-blockers and the second group (group 2) are participants not-taking beta-blockers.

ELIGIBILITY:
Inclusion Criteria:

- Patients taking and not taking beta-blockers

Exclusion Criteria:

* Participants with heat and neck or esophageal cancer
* Participants with stroke or neurological disease
* Participants with central nervous system disease
* Participants with concomitant treatment with Angiotensin converting enzyme inhibitors (ACEI), Angiotensin II receptor antagonists (ARA-II), Antipsychotics, Dopamine agonists, Capsaicine.
* Participants with severe clinical signs of aspiration, including oxygen desaturation ≥3%.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All population.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-11-25 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Substance P levels | 1 year
  In blood and saliva

CONTACTS AND LOCATIONS:
Overall Officials: Marta Miarons, Principal Investigator — Mataró Hospital
Locations (1):
- Mataró Hospital, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided